CLINICAL TRIAL: NCT04968366
Title: Phase I Clinical Study of Safety & Efficacy of DC Vaccine and TMZ for the Treatment of Newly-diagnosed Glioblastoma After Surgery
Brief Title: Safety & Efficacy of DC Vaccine and TMZ for the Treatment of Newly-diagnosed Glioblastoma After Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: ZhongSheng BioTech Inc. (Unknown)
Responsible Party: Principal Investigator, Yang Zhang, Chief Neurosurgeon, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY 2021-021-02
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma Multiforme of Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DC vaccine group (Experimental): Subjects will receive five to eight doses of the DC vaccine through i.d. injection into regions near to the groin and axillary during they receive TMZ adjuvant chemotherapy
  Interventions: Biological: Autologous dendritic cells pulsed with multiple neoantigen peptides.; Drug: Temozolomide adjuvant chemotherapy

INTERVENTIONS:
Biological: Autologous dendritic cells pulsed with multiple neoantigen peptides. — Each dosage of Dendritic Cells (DC) vaccine contains 2-10 million DC cells, loaded with 5-20 tumor neoantigen peptides. DC vaccine will be administered (i.d) around lymph nodes of the groin and Axillary at 2nd, 3rd, 4th, 7th and 11th week after the completion of concurrent Temozolomide chemoradiation. After 5 injections, the investigator will review subject's tolerance and compliance; and, decide whether to administer more DC vaccines up to 8 injections. For certain patients with good tolerance and clinical response of the DC vaccine, peripheral blood is extracted after completion of Temozolomide adjuvant chemotherapy to assess the patient's immune response. According to the result, investigators will decide whether to perform 1-2 more treatment cycles (5-8 injections/cycle) to strengthen the effectiveness
Drug: Temozolomide adjuvant chemotherapy — Temozolomide is administered as the standard-of-care adjuvant chemotherapy, in combination with the DC vaccines to treat the enrolled patients.
  Other Names: the standard-of-care adjuvant chemotherapy for GBM patients

SUMMARY:
This is a single-center, single-arm phase I study to determine the safety and preliminary efficacy of autologous dendritic cells (DCs) loaded with multiple tumor neoantigen peptides administered as a cancer-treatment vaccine to treat adult postoperative patients with newly-diagnosed glioblastoma, in combination with the standard-of-care Temozolomide (TMZ) chemotherapy.

DETAILED DESCRIPTION:
This is a single-center, single-arm phase I study to determine the safety and preliminary efficacy of autologous dendritic cells (DCs) loaded with multiple tumor neoantigen peptides administered as a cancer-treatment vaccination for the treatment of newly-diagnosed glioblastoma (GBM). The subjects are adult GBM patients who have undergone surgical resection. After the completion of TMZ concurrent chemoradiation, and, during conventional adjuvant TMZ chemotherapy, subjects will receive autologous DC vaccine treatments as scheduled. Ten subjects will be enrolled. The autologous genetic-modification-free DC cells will be loaded with multiple tumor neoantigen peptides and administered (i.d) to subjects. After 5 injections, the investigator will review subject's tolerance and compliance, and decide whether or not to administer more DC vaccines up to 8 injections. For certain patients with good tolerance and clinical response of the DC vaccine, peripheral blood is extracted after completion of TMZ adjuvant chemotherapy to assess patient's immune response. According to the result, investigators will be decided whether to perform more 1-2 treatment cycles (5-8 infections/cycle) to strengthen the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years (including 18 and 75 years old);
2. Newly-diagnosed glioblastoma confirmed by histopathological exams;
3. IDH1- and IDH2-wild-type gliomas;
4. Extent of resection of enhancing lesions > 90%;
5. Karnofsky Performance Score(KPS) ≥ 60%;
6. Adequate organ functions:

The absolute value of white blood cells ≥ 2.5×10 9/L; Hemoglobin levels> 100 g/L; Platelet counts > 100×109/L; Levels of Alanine aminotransferase, aspartate aminotransferase <2.5 x ULN; Serum creatinine levels <1.5 x ULN.

Exclusion Criteria:

1. Subjects with any other active malignancy;
2. Subjects received the placement of Carmustine implants within 6 months before the inclusion;
3. Subjects with active HBC, HCV or HIV infection;
4. Subjects with grade 2 -3 hypertension or uncontrolled hypertension;
5. Subjects with severe cardio- or cerebro- vascular diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, etc.;
6. Subjects with uncontrolled autoimmune diseases such as hemolytic anemia, psoriasis and rheumatoid arthritis, etc.;
7. Subjects with severe or uncontrolled psychiatric diseases or condition that could increase adverse events or interfere the evaluation of outcomes;
8. Subjects receiving immunosuppressants after organ transplantation;
9. Within four weeks before the DC vaccinations, subjects receiving systemic administration of steroids with dosage more than 10mg/d prednisone or the equivalent doses of other steroids ( not including inhaled corticosteroid);
10. Subjects with unstable pulmonary embolism, deep venous embolism, or other major arterial and venous thromboembolic events that occur within 30 days before the enrollment; receiving ongoing anticoagulant therapy;
11. Subjects in pregnancy or breastfeeding, or those who plan to become pregnant during treatment or within 2 months after the end of treatment;
12. Within the 14 days before enrollment, subjects with active infections or uncontrolled infections that require systemic antibiotic treatment (except for simple urinary tract infections or upper respiratory tract infections);
13. Subjects who have received other vaccine therapies or gene-modified cell therapy before enrollment;
14. Subjects with number of the predicted neoantigen peptides less than 5;
15. Subjects with other conditions that would interfere trial participation at the investigator's discretion;
16. Subjects with medical conditions that affect signing the written informed consent or complying with the research procedures; or patients who are unwilling or unable to comply with the research procedures;
17. Subjects who participated or are participating in other clinical trials within 4 weeks before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) | All the AEs were recorded from the first shot to 8 weeks after the last shot.
  AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Proportions of patients with positive peripheral tumor specific immune response after the DC vaccinations | start from the inclusion timepoint to one week after the last injection.
  The peripheral tumor specific immune response is measured by the IFN-γ release ELISPOT assay, using the peripheral blood mononuclear cells (PBMCs) that are collected before the vaccine injection (baseline), one week after the 3r, 5th and the last injection, respectively. The positive response is defined as "≥ 55 spot-forming cells in each million PBMCs" or "number of spot-forming cells increase by 3-fold after the DC vaccination compared with the baseline".
Progression-free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  months from the date of surgery to tumor recurrence or progression
Overall survival | From date of surgery until the date of death from any cause, assessed up to 60 months
  months from the date of surgery to death
Rate of the patients who survive for more than one year after surgery in all the included patients who receive the DC vaccine | From date of surgery until one year after surgery
  One-year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, Dr., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No